CLINICAL TRIAL: NCT06407947
Title: Exploratory Clinical Trial of the Safety and Efficacy of CT071 Injection in Patients With High Risk Newly Diagnosed Multiple Myeloma
Brief Title: Study of CT071 Injection in High Risk Newly Diagnosed Multiple Myeloma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT071-CG7002
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Chimeric antigen receptor modified T cells
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chimeric antigen receptor modified T cells Infusion (Experimental): Chimeric antigen receptor modified T cells chimeric antigen receptor T cells
  Interventions: Drug: Chimeric antigen receptor modified T cells Infusion

INTERVENTIONS:
Drug: Chimeric antigen receptor modified T cells Infusion — chimeric antigen receptor T cells
  Other Names: Single Group Assignment

SUMMARY:
This trial is a single-arm, single-center, open-label clinical trial to evaluate the safety, efficacy, and metabolism kinetics of CT071 in patients with high-risk newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
This trial is a single-arm, single-center, open-label clinical trial to evaluate the safety, efficacy, and metabolism kinetics of CT071 in patients with high-risk newly diagnosed multiple myeloma (HRNDMM).

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be enrolled:

1.Volunteer to participate in the clinical trial; the participants themselves fully understand and are informed of this study, and sign the informed consent form and are willing to follow and able to complete all trial procedures;

2.Age ≥ 18 years, male or female;

3.Participants must have newly diagnosed with multiple myeloma according to International Myeloma Working Group diagnostic criteria 2014 ;

4.Measurable disease based on at least one of the following parameters (International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma 2016); the values for these parameters obtained up to 60 days prior to signing the Informed Consent Form including the results at the time of diagnosis may be used.

1. Serum M-protein ≥ 1.0 g/dL;
2. Urine M-protein ≥ 200 mg/24 hr;
3. Serum free light chain (FLC): involved FLC level ≥ 10 mg/dL (100 mg/L) provided serum FLC ratio is abnormal.

   5.Known to have the following high risk factors, i.e. At least one of the following conditions is met:

   1)Meet any one or more of the cytogenetic criteria: del (17p); t (4; 14); t (14; 16); t (14; 20); 1q21 amplification ≥ 4 copies; 2)R-ISS stage 3; R2-ISS stages 3 and 4; 3)Presence of soft tissue extramedullary plasmacytoma 4)2%-5% in peripheral plasma cells;

   6.Eastern Cooperative Oncology Group (ECOG) score 0-2;

   7.Participants should meet the following test results (repeat tests are allowed):

   1)Hematology: Absolute neutrophil (ANC) count ≥ 1.0 × 109/L; Platelet (PLT) ≥ 50 × 109/L; Hemoglobin (Hb) ≥ 7.5 g/dL; 2)Blood chemistry: Endogenous creatinine clearance ≥ 40 mL/min (see Appendix 1 using the Cockcroft-Gault formula); Alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN), aspartate aminotransferase (AST) ≤ 2.5 × ULN, total bilirubin ≤ 1.5 × ULN; 3)International normalized ratio (INR), or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN.

   8.Venous access required for collection can be established and there is no contraindication for cell collection.

   9.Females of childbearing potential (WOCBP) must have a negative serum pregnancy test at screening and must be willing to use effective and reliable contraception for at least 12 months after CT071 infusion.

   10.A male participant, if sexually active with a female of childbearing potential, is willing to use a highly effective and reliable method of contraception for 1 year after receiving trial treatment. All male participants absolutely refrain from donating sperm during the trial and for 1 year after receiving trial treatment.

   Exclusion Criteria:

   Participants were not enrolled in the trial if they met any of the following criteria:
   1. Patients with non-secretory MM.
   2. Prior treatment for MM other than up to 2 cycles of (bortezomib, lenalidomide, dexamethasone) for induction, including but not limited to cytotoxic therapy, proteasome inhibitors, immunomodulators, targeted therapy, radiotherapy (patients are eligible for this trial if the radiation field covers ≤ 5% bone marrow reserve regardless of the end date of radiotherapy), epigenetic therapy, etc.
   3. Pregnant or lactating females.
   4. Patients with severe mental disorders or altered mental status, history of central nervous system disease, such as epilepsy, intracranial hemorrhage, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, memory impairment, spinal cord compression, psychiatric disease or any disease involving the central nervous system, or suspected central nervous system (CNS) metastasis, or any autoimmune disease involving the CNS, with or suspected CNS infiltration.
   5. Participants had other malignancies, including the following that were considered to have been successfully treated: non-metastatic basal cell or squamous cell skin cancer, non-metastatic prostate cancer, carcinoma in situ of the breast or cervix, and non-muscle invasive bladder cancer.
   6. Active autoimmune disease that results in end organ damage or requires systemic immunosuppressive/systemic disease modifying drugs, including but not limited to Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus and other patients requiring long-term immunosuppressive therapy.
   7. Have any uncontrolled active infection (defined as exhibiting persistent signs or symptoms associated with infection that do not improve despite appropriate anti-infective therapy), or other serious active viral, bacterial, or uncontrolled systemic fungal infection. I
   8. Positive test results for biomarkers of any of the following pathogenic microorganisms: human immunodeficiency virus (HIV) antibody, Treponema pallidum antibody (TPPA), hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) (core antigen [HBcAb] positive must have DNA copies below the lower limit of normal).
   9. Vaccination with live attenuated vaccine or mRNA vaccine within 8 weeks and inactivated vaccine within 4 weeks prior to screening.
   10. Patients who are allergic or intolerant to lymphodpletion drugs, tocilizumab, or allergic to the ingredients of CT071 cell infusion preparation (DMSO); Or previous history of other severe allergies, such as anaphylactic shock.
   11. Clinically significant cardiac abnormalities, including but not limited to:

   1)Uncontrolled congestive heart failure (New York Heart Association Class III or IV heart failure, see Appendix 3); 2)Myocardial infarction, coronary artery bypass grafting or unstable angina within 6 months prior to apheresis; 3)History of clinically significant uncontrolled cardiac arrhythmias such as ventricular arrhythmias; 4)History of severe non-ischemic cardiomyopathy; 5)Left ventricular ejection fraction (LVEF) < 50%, diagnosed by echocardiography, without clinically significant ECG abnormalities; 6)Other heart disease that, in the opinion of the investigator, may jeopardize the health of the participant when participating in this clinical trial.

   12.Participants with known or suspected chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% of the predicted normal value of spirometry, or other lung disease that, in the judgment of the investigator, significantly affects lung function or affects the safety of the participant, such as asthma, interstitial lung disease, diffuse lung disease, pulmonary infection, pulmonary embolism, etc.

   13.No need for supplemental oxygen for maintenance and oxygen saturation < 92% in room air.

   14.Participant has a history of stroke or seizure within 6 months prior to the screening period.

   15.Has had major surgery before screening, or is planned to undergo major surgery after the trial treatment (excluding cataract and other surgery under local anesthesia). The investigator must discuss with the sponsor to determine whether a surgery is major surgery before enrolling the participant in the trial.

   16.The participant has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) v5.0 ≤ Grade 1 from toxicities attributable to previous treatments, except for alopecia, peripheral neuropathy, and other events that, in the judgment of the investigator, are unlikely to result in lymphodepletion or cumulative toxicities of CT071 treatment; 17.Other conditions considered inappropriate for participation in this clinical trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2027-06-03 (Estimated); Study Completion 2027-06-03 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) after CT071 infusion | From first dose of study drug administration to end of treatment (up to 24 months)
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), with the exception of cytokine release syndrome (CRS), and immune effector cell-associated neurotoxicity syndrome (ICANS).
Overall response rate (ORR) | From first dose of study drug administration to end of treatment (up to 24 months)
  ORR defined as proportion of patients achieving partial response or better based on International Myeloma Working Group defined response criteria
Recommended Phase II Dose of CT071 in patients with high-risk newly diagnosed multiple myeloma | Assessed from the date of first dose of study treatment until 28 days
  Evaluate Dose limited toxicity and adverse events after CT071 infusion

SECONDARY OUTCOMES:
Minimal residual disease (MRD) negative rate | From first dose of study drug administration to end of treatment (up to 24 months)
  Minimal residual disease (MRD) negative rate is defined as the proportion of patients with Very good partial response or better who achieved 10-5 sensitivity of nucleated cell
Complete response/stringent complete response (CR/sCR) rate | From first dose of study drug administration to end of treatment (up to 24 months)
  Rate of complete response/stringent complete response (CR/sCR) defined as proportion of patients achieving CR or better based on International Myeloma Working Group defined response criteria
Duration of response (DOR) | From first dose of study drug administration to end of treatment (up to 24 months)
  DOR is defined as the time from first achieving partial response or better to confirmed disease progression or death from any cause
Progression-free survival (PFS) | From first dose of study drug administration to end of treatment (up to 24 months)
  PFS defined as the time from the date of apheresis of the subject to the first assessment of confirmed disease progression or death from any cause according to International Myeloma Working Group 2016 criteria, whichever occurs first
Time to response (TTR) | From first dose of study drug administration to end of treatment (up to 24 months)
  TTR defined as the time from the date of apheresis to the date of initial assessment of Partial response or better according to International Myeloma Working Group 2016 criteria
Time to best response (TTBR) as assessed by the investigator | From first dose of study drug administration to end of treatment (up to 24 months)
  TTBR defined as the time from the date of apheresis to the date of assessment with a best response according to International Myeloma Working Group 2016 criteria
Overall survival (OS) | From first dose of study drug administration to end of treatment (up to 24 months)
  OS defined as the time from the date of apheresis of the subject to death from any cause
Peak Plasma Concentration (Cmax) of CAR T cells | From first dose of study drug administration to end of treatment (up to 24 months)
  time to Peak Plasma Concentration (Cmax)
Presence of anti-CT071 antibodies | From first dose of study drug administration to end of treatment (up to 24 months)
  Anti-drug antibody positive rate
Duration of MRD negativity | From first dose of study drug administration to end of treatment (up to 24 months)
  Sustain MRD negative month
Cytokines in the peripheral blood after CT071 infusion | From first dose of study drug administration to end of treatment (up to 24 months)
  Serum concentrations of granulocyte-macrophage colony stimulating factor (GM-CSF) interleukin (IL)-6, IL-10, interferon gamma (IFN-γ) and tumor necrosis factor (TNF),after CT071 infusion
Immune-related proteins after CT071 infusion | From first dose of study drug administration to end of treatment (up to 24 months)
  Serum concentrations of C-reactive protein (CRP),etc.
Markers | From first dose of study drug administration to end of treatment (up to 24 months)
  Expresion of soluble GPRC5D (sGPRC5D)
Area under the plasma concentration versus time curve (AUC) of CART cells | From first dose of study drug administration to end of treatment (up to 24 months)
  Area under the plasma concentration versus time curve (AUC)
Level of CAR-T Cell Expansion persistence | From first dose of study drug administration to end of treatment (up to 24 months)
  Levels of cell expansion persistence via monitoring CAR-T positive cell counts and CAR transgene level will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Du, Shanghai, Shanghai Municipality, China